CLINICAL TRIAL: NCT06186622
Title: A Drug-Drug Interaction Study to Assess the Effect of Orforglipron on the Pharmacokinetics of Digoxin, Simvastatin, Rosuvastatin, Acetaminophen, and Midazolam in Healthy Overweight and Obese Participants
Brief Title: A Drug-Drug Interaction Study of Orforglipron (LY3502970) in Healthy Overweight and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18631; J2A-MC-GZPG (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Obese; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron; Simvastatin; Digoxin; Rosuvastatin Calcium; Acetaminophen; Midazolam; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Part 1) (Experimental): Participants will receive Orforglipron capsule and tablet formulation with Simvastatin, Digoxin, Rosuvastatin, Acetaminophen, Midazolam and Sodium Bicarbonate administered orally.
  Interventions: Drug: Orforglipron; Drug: Simvastatin; Drug: Digoxin; Drug: Rosuvastatin; Drug: Acetaminophen; Drug: Midazolam; Drug: Sodium Bicarbonate
- Orforglipron (Part 2) (Experimental): Participants will receive Orforglipron capsule and tablet formulation with Simvastatin, Digoxin and Sodium Bicarbonate administered orally.
  Interventions: Drug: Orforglipron; Drug: Simvastatin; Drug: Digoxin; Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
Drug: Simvastatin — Administered orally.
Drug: Digoxin — Administered orally.
Drug: Rosuvastatin — Administered orally.
  Arms: Orforglipron (Part 1)
Drug: Acetaminophen — Administered orally.
  Arms: Orforglipron (Part 1)
Drug: Midazolam — Administered orally.
  Arms: Orforglipron (Part 1)
Drug: Sodium Bicarbonate — Administered orally.

SUMMARY:
The main purpose of this study is to determine effect of orforglipron capsule formulation on the amount of digoxin, rosuvastatin, acetaminophen, midazolam, and simvastatin (each given alone and together with orforglipron) that enters the bloodstream and how long it takes the body to eliminate them when administered orally in healthy overweight and obese participants. In addition, the effect of the orforglipron tablet on the amount of simvastatin that enters the bloodstream and how long it takes the body to eliminate it will be evaluated.

The study will also assess the effect of sodium bicarbonate when administered alone with simvastatin versus orforglipron capsule containing sodium bicarbonate administered with simvastatin. The safety and tolerability of orforglipron and information about any side effects experienced will be collected.

Study will be conducted in two parts, with part 1 and 2 lasting up to approximately 23 and 24 weeks each, including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical history and physical examination.
* Have body mass index (BMI) equal to or greater than 27 kilograms per meter squared (kg/m²), inclusive, at screening.
* Have an estimated glomerular filtration rate equal to or greater than 60 milliliters per minute (mL/min).
* Males and females who agree to follow contraceptive requirements, or women not of childbearing potential (WNOCBP).
* Have venous access sufficient to allow for blood sampling.

Exclusion Criteria:

* Have any type of diabetes with hemoglobin A1c (HbA1c) level of 6.5 percent (%) or greater.
* Have significant history of or currently have Major Depressive Disorder or psychiatric disorder within the last 2 years.
* Obesity induced by other endocrine disorders, such as Cushing's syndrome or Prader-Willi syndrome.
* Have known clinically significant gastric emptying abnormality.
* Have undergone bariatric surgery (for example: Lap-Band, Gastric Bypass)
* Have a known self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or any form of thyroid cancer.
* Have an abnormal 12-lead electrocardiogram (ECG) at screening.
* Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drug.
* Participants must not be currently participating in or completed a clinical trial within the last 90 days.
* Have a known allergy or hypersensitivity to midazolam, simvastatin, rosuvastatin, or digoxin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC [0-∞]) of Simvastatin and simvastatin acid following simultaneous administration of Orforglipron capsule formulation | Predose up to 24 hours postdose
  PK: AUC [0-∞] of Simvastatin and simvastatin acid following simultaneous administration of Orforglipron capsule formulation
PK: AUC [0-∞] of Simvastatin and simvastatin acid following staggered administration of Orforglipron capsule formulation | Predose up to 24 hours postdose
PK: AUC [0-∞] of Simvastatin and simvastatin acid after sodium bicarbonate coadministration | Predose up to 24 hours postdose
PK: AUC [0-∞] of Digoxin | Predose up to 120 hours postdose
PK: AUC [0-∞] of Rosuvastatin | Predose up to 72 hours postdose
PK: AUC [0-∞] of Acetaminophen | Predose up to 24 hours postdose
PK: AUC [0-∞] of Midazolam and 1'-hydroxymidazolam | Predose up to 24 hours postdose
PK: Maximum Observed Concentration (Cmax) of Simvastatin and simvastatin acid following simultaneous administration of Orforglipron capsule formulation | Predose up to 24 hours postdose
  PK: Cmax of Simvastatin and simvastatin acid following simultaneous administration of Orforglipron capsule formulation
PK: Cmax of Simvastatin and simvastatin acid following staggered administration of Orforglipron capsule formulation | Predose up to 24 hours postdose
PK: Cmax of Simvastatin and simvastatin acid after sodium bicarbonate coadministration | Predose up to 24 hours postdose
PK: Cmax of Digoxin | Predose up to 120 hours postdose
PK: Cmax of Rosuvastatin | Predose up to 72 hours postdose
PK: Cmax of Acetaminophen | Predose up to 24 hours postdose
PK: Cmax of Midazolam and 1'-hydroxymidazolam | Predose up to 24 hours postdose

SECONDARY OUTCOMES:
PK: AUC [0-∞] of Simvastatin and simvastatin acid after administrating Orforglipron tablet formulation | Predose up to 24 hours postdose
PK: Cmax of Simvastatin and simvastatin acid after administrating Orforglipron tablet formulation | Predose up to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Fortrea Clinical Research Unit Inc., Daytona Beach, Florida
  - Fortrea Clinical Research Unit Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No